CLINICAL TRIAL: NCT01511198
Title: NNC 90-1170 Dose-response, Efficacy and Safety: A 12-week Randomized, Multicenter, Doubleblind, Double-dummy, Parallel-group Study of Metformin and Five Doses of NNC 90-1170 in Previously-treated OHA Monotherapy Obese Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Metformin and Liraglutide in Obese Subjects With Type 2 Diabetes Previously Treated With an Oral Hypoglycemic Agent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-2072
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 0.045 mg (Experimental)
  Interventions: Drug: liraglutide
- 0.225 mg (Experimental)
  Interventions: Drug: liraglutide
- 0.45 mg (Experimental)
  Interventions: Drug: liraglutide
- 0.60 mg (Experimental)
  Interventions: Drug: liraglutide
- 0.75 mg (Experimental)
  Interventions: Drug: liraglutide
- Met (Active Comparator)
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: liraglutide — Injected subcutaneously once daily
  Other Names: NNC 90-1170
  Arms: 0.045 mg; 0.225 mg; 0.45 mg; 0.60 mg; 0.75 mg
Drug: metformin — 1000 mg twice daily, administered orally
  Arms: Met

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to determine the dose-response relationship for body weight and five escalating doses of NNC 90-1170 (liraglutide) in subjects with type 2 diabetes previously treated with an oral hypoglycemic agent (OHA).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic
* Treated with OHA (oral hypoglycaemic agent monotherapy for at least 3 months. Prior use of metformin is allowed
* Body Mass Index (BMI) between 27.0-42.0 kg/m^2 (inclusive)
* HbA1c maximum 10% based on analysis from central laboratory

Exclusion Criteria:

* Cardiac problems
* Uncontrolled treated/untreated hypertension
* Proliferative retinopathy or known autonomic neuropathy
* Recurrent severe hypoglycemia as judged by the investigator
* Known or suspected allergy to trial product or related products
* Use of any drug (except for OHAs), which in the investigators opinion could interfere with the glucose level or body weight or any contraindication to metformin use or intolerance to metformin 1000 mg (prior to trial entry or during run-in period). Stable doses, for 3 months or greater, of thyroid hormone replacement are allowed
* Known or suspected abuse of alcohol or narcotics
* Current treatment with thiazolidinediones or chronic daily use of insulin (more than 7 days) within three months in the absence of intercurrent illness
* TSH (thyroid stimulating hormone) below 0.2 or above 15 U/mL
* Type 1 or other specific causes of diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2001-02; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Body weight

SECONDARY OUTCOMES:
FPG (fasting plasma glucose)
HbA1c (glycosylated haemoglobin)
Fructosamine
Lipids
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (35):
- United States (35):
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Carlisle, Arkansas
  - Novo Nordisk Investigational Site, Jonesboro, Arkansas
  - Novo Nordisk Investigational Site, Alhambra, California
  - Novo Nordisk Investigational Site, Mission Viejo, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Trumbull, Connecticut
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Titusville, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Duluth, Minnesota
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, North Plainfield, New Jersey
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Edmonds, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Tacoma, Washington
  - Novo Nordisk Investigational Site, Charleston, West Virginia

REFERENCES:
- [Result] Feinglos MN, Saad MF, Pi-Sunyer FX, An B, Santiago O; Liraglutide Dose-Response Study Group. Effects of liraglutide (NN2211), a long-acting GLP-1 analogue, on glycaemic control and bodyweight in subjects with Type 2 diabetes. Diabet Med. 2005 Aug;22(8):1016-23. doi: 10.1111/j.1464-5491.2005.01567.x. PMID 16026367
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com